CLINICAL TRIAL: NCT04815863
Title: A Comparison of Somatic Symptom Among Elderly and Non-elderly in Chinese Community-Dwelling People
Brief Title: Assessment of Somatic Symptom in Chinese Community-Dwelling People
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SSSCN202011
Record Dates: First submitted 2020-12-06; First posted 2021-03-25 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Somatization Disorder
Keywords: somatic symptom disorder; Somatic Symptom Scale-China; elderly
MeSH Terms: conditions — Somatoform Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly: Over 60 years old
  Interventions: Diagnostic Test: Assessment of somatic symptom disorder with SSS-CN; Diagnostic Test: Assessment of depressive symptoms disorder with PHQ-9; Diagnostic Test: Assessment of anxiety disorder with GAD-7
- Non-Elderly: Under 60 years old
  Interventions: Diagnostic Test: Assessment of somatic symptom disorder with SSS-CN; Diagnostic Test: Assessment of depressive symptoms disorder with PHQ-9; Diagnostic Test: Assessment of anxiety disorder with GAD-7

INTERVENTIONS:
Diagnostic Test: Assessment of somatic symptom disorder with SSS-CN — SSS-CN questionnaire is used to assess the presence and severity of the somatic symptoms
Diagnostic Test: Assessment of depressive symptoms disorder with PHQ-9 — PHQ-9 questionnaire is used to assess the presence and severity of the depressive symptoms
Diagnostic Test: Assessment of anxiety disorder with GAD-7 — GAD-7 questionnaire is used to assess the presence and severity of the anxiety disorder

SUMMARY:
With the rapid aging and worsening psychological problems worldwide, the special focus on somatic symptom and other psychological diseases of the older population is needed. However, there is no research comparing the incidence of somatic symptom between elderly and non-elderly, and clinical relevance with somatic symptom is uncertain. The study aims to clarify the prevalence of somatic symptom, depression and anxiety disorders in China, to compare physical and psychological difference between the elderly and non-elderly and to explore risk factors for somatic symptom in the elderly.

DETAILED DESCRIPTION:
With the steadily increasing of life expectancy, the aging people is expected to 2 billion by 2050, which brings the deeper demand on the quality of life improvement. The psychological problems is an important factor affecting the quality of life. As reported, 73.6% of urban residents were with mental sub-health, indicating that psychological problem has grown into inevitable issues in hindering healthy development. The elderly, compared with the non-elderly, have unique social and biological characteristics, so psychological problem of the older population deserves special focus. Literatures have investigated aged people with depression or anxiety disorder, but somatic symptom in elderly have rarely been addressed. Somatic symptom disorder prevalence in elderly in European ranged from 0-13.5%. However, there is no research comparing the incidence of somatic symptom, anxiety and depression between elderly and non-elderly and revealing the prevalence of somatic symptom under Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria.

Investigators use Somatic Symptom Scale-China (SSS-CN) questionnaire to assess the presence and severity of the symptoms. Patient Heath Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder Screener (GAD-7) are used to evaluate depression and anxiety disorder respectively. The study aims to clarify the prevalence of somatic symptom, depression and anxiety disorders in China, to compare physical and psychological difference between the elderly and non-elderly and to explore risk factors for somatic symptom in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. voluntary participants and gave written consent to participates the study;
2. undertook SSS-CN questionnaire, PHQ-9 and GAD questionnaires；

Exclusion Criteria:

1. patients who have lost their self-assessed abilities or refuse to participate ;
2. patient with cancer and central nervous system disease;
3. patients who have been previously confirmed serious mental disorders, mental retardation or dementia.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects are enrolled between March 2019 and June 2019 in 105 representative community health service institutions in Shanghai, China.
Sampling Method: Probability Sample
Enrollment: 9110 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiantong University
Locations (2):
- China (2):
  - Renji Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elderly | Non-Elderly
Started | 6874 | 2236
Completed | 6814 | 2206
Not Completed | 60 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderly | Non-Elderly | Total
Number analyzed (Participants) | 6814 | 2206 | 9020
Age, Customized [Count of Participants; unit: Participants]
  18-59 | 0 | 2206 | 2206
  ≥60 | 6814 | 0 | 6814
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Information missing
  Participants
    number analyzed (Participants) | 6798 | 2202 | 9000
    Female | 2567 | 693 | 3260
    Male | 4231 | 1509 | 5740
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 6814 | 2206 | 9020
Education [Count of Participants; unit: Participants] — Population: Information missing
  Participants
    number analyzed (Participants) | 6798 | 2202 | 9000
    Middle School and below | 3481 | 670 | 4151
    High school | 2010 | 617 | 2627
    College | 1262 | 859 | 2121
    Master and above | 45 | 56 | 101
Hypertension [Count of Participants; unit: Participants]
  Yes | 3621 | 409 | 4030
  No | 3193 | 1797 | 4990
Diabetes mellitus [Count of Participants; unit: Participants]
  Yes | 1731 | 190 | 1921
  No | 5083 | 2016 | 7099
Cardio/Cerebrovascular disease [Count of Participants; unit: Participants]
  Yes | 1910 | 154 | 2064
  No | 4904 | 2052 | 6956
Other disease [Count of Participants; unit: Participants]
  Yes | 123 | 29 | 152
  No | 6691 | 2177 | 8868
Surgery [Count of Participants; unit: Participants]
  Yes | 75 | 4 | 79
  No | 6739 | 2202 | 8941
Antipsychotics [Count of Participants; unit: Participants]
  Yes | 154 | 8 | 162
  No | 6660 | 2198 | 8858
Marital status [Count of Participants; unit: Participants] — Population: Information missing
  Participants
    number analyzed (Participants) | 6798 | 2202 | 9000
    Never married | 307 | 172 | 479
    Married | 5868 | 1842 | 7710
    Divorced | 90 | 23 | 113
    Widowed | 533 | 165 | 698

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Somatic Symptoms Disorder
Description: The scores of Somatic Symptom Scale-China (SSS-CN) questionnaire were recorded. The score higher than 20 was taken as somatic symptom disorder. Percentage of somatic symptom disorder in elderly and in non-elderly were analyzed.
Time Frame: Within 24 hours of the questionnaire completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Elderly | Non-Elderly
Number analyzed (Participants) | 6814 | 2206
Participants
  Yes | 4307 | 1000
  No | 2507 | 1206

2. Other Pre Specified Outcome: Number of Participants With Somatic Symptoms Disorder Accompanied With Anxiety
Description: anxiety disorder were assessed by Generalized Anxiety Disorder-7 (GAD-7). The percentage of anxiety disorder among the participants with somatic symptoms disorder were analyzed.
Time Frame: Within 24 hours of the questionnaire completion.
Measure: Count of Participants; unit: Participants
Groups:
- Elderly With SSD: Elderly with SSD
- Non-Elderly With SSD: Non-Elderly with SSD
Arm/Group | Elderly With SSD | Non-Elderly With SSD
Number analyzed (Participants) | 4307 | 1000
Participants
  With anxiety disorder | 709 | 233
  Without anxiety disorder | 3598 | 767

3. Other Pre Specified Outcome: Number of Participants With Somatic Symptoms Disorder Accompanied With Depression
Description: Depressive disorder were assessed by Patient Health Questionnaire-9 (PHQ-9). The percentage of depressive disorder among the participants with somatic symptoms disorder were analyzed.
Time Frame: Within 24 hours of the questionnaire completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Elderly With SSD | Non-Elderly With SSD
Number analyzed (Participants) | 4307 | 1000
Participants
  With depressive disorder | 1104 | 306
  Without depressive disorder | 3203 | 694

ADVERSE EVENTS:
Time Frame: During the 1-day window allocated for questionnaire administration and medical history collection.
Description: Not availale.
Arm/Group | Elderly | Non-Elderly
All-Cause Mortality (participants affected / at risk) | 0/6814 | 0/2206
Serious Adverse Events (participants affected / at risk) | 0/6814 | 0/2206
Other Adverse Events (participants affected / at risk) | 0/6814 | 0/2206

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT04815863/Prot_SAP_000.pdf